CLINICAL TRIAL: NCT05591729
Title: Effect of Pilates on Balance and Spinal Curvature In Upper Crossed Syndrome
Acronym: UCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam omran Grase, principle investigator mariam omran grase, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T/012/003992
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Postural; Defect
Keywords: pilates exercise; upper cross syndrome; balance; spinal curvature
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus; Spinal Curvatures | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: pilates exercise and postural correction group
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercise (Experimental): pilates exercise will be received twice a week for four weeks
  Interventions: Other: Pilates exercises; Other: postural correction exercise
- postural correction exercise (Active Comparator): postural correction exercises will be received twice a week for four weeks
  Interventions: Other: postural correction exercise

INTERVENTIONS:
Other: Pilates exercises — Each Pilates session will last for one hour. The subjects will be taught the 5 key elements of Pilates (lateral costal breathing, centering which is a neutral position of the lumbar spine with activation of the core muscles, ribcage placement, shoulder blade placement and neutral position of the cervical spine with slight upper cervical flexion at the craniocervical junction). A pilates exercise program will consist of 11 levels of treatment program.
  Arms: Pilates exercise
Other: postural correction exercise — the patients will receive postural correction exercises, stretches, and exercises to the pectoralis major, elevator scapulae, upper trapezius, serratus anterior, rhomboids, and deep neck flexors. The stretches included sitting chair stretches, Brugger's, wall angels, and doorway stretches. The exercises included push-up-plus, head-neck-retraction, and Kibler squeeze

SUMMARY:
The study will be conducted to investigate the effect of Pilates exercise on spinal curvature and balance in patients with the upper cross syndrome. .

DETAILED DESCRIPTION:
Upper crossed syndrome (UCS) is the most common postural dysfunction in the musculature of the shoulder girdle /cervicothoracic region, which creates joint dysfunction, particularly at the atlanto-occipital joint, cervicothoracic joint C4-C5 segment, glenohumeral joint and T4-T5 segment. Pilates is designed as a program that will work with other exercise programs to strengthen, rebalance and realign the body. Pilates trains individuals to identify their own musculoskeletal strengths and weaknesses and equips them with the knowledge to correct and rebalance their entire body mechanics (Worth,2004) thus, the focus is also placed on improving personal body awareness which further decreases the risks of strain or injury that can occur with imbalances. forty patients with UCS will be allocated randomly into two groups; one experimental group will receive pilates exercise and postural correction twice a week for four weeks, and the control group will receive postural correction exercise along twice a week for four weeks

ELIGIBILITY:
Inclusion Criteria:

* The patient's age ranged from 17 to 22 years
* Body mass index between 20-25 kg/m2
* The participants are diagnosed with upper cross syndrome
* Patients with normal cognitive aspects willing and able to participate in a program safely

Exclusion Criteria:

* The participants have experienced any recent trauma (within 3 months of the initial consultation)
* The participant's primary complaint is that of headaches or facial pain.
* Contra-indications to pilates are found pregnancy, hypertension, osteoporosis, and spinal tumors.
* Participants have any sort of structural abnormality in upper and middle back e.g., Scoliosis, or had a positive Adams test.
* Participants who are taking anti-inflammatory or muscle relaxant medication had to have a three-day "wash out" period before participating in the study

Ages: 17 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
spinal curvature | up to four weeks
  spinal mouse will be used to assess thoracic spine curvature. Total angle of the thoracic spine is 41-44 degree.
balance | up to four weeks
  balance will be measured by Biodex balance system

SECONDARY OUTCOMES:
craniovertebral angle | up to four weeks
  craniovertebral angle will be measured by photogrammetric method
pain intensity | up to four weeks
  pain will be measured by visual analogue scale
neck function | up to four weeks
  neck function will be measured by Arabic neck disability index.. It consisting of 10 items with six choices. There is no disability for scores from 0 to 4; 5-14 is mild; 15-24 is moderate; 25-34 is severe, and finally more than 34 is a complete disability.
shoulder posture | up to four weeks
  The shoulder's rounded position will be measured by tap measurement. the patients will be in supine and the therapist measure the distance from their shoulder to the plinth using tape measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy Cairo, Giza, Egypt